CLINICAL TRIAL: NCT04857489
Title: Deficient T Regulatory Cell (Treg) Function in Patients With Relapsing Remitting Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 19S.016
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Relapse Remitting Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Relapse Remitting Multiple Sclerosis: Blood sample
- Healthy Controls: Blood Sample

SUMMARY:
The purpose of this research is to find out how the T regulatory (Treg) cells control autoimmune response in multiple sclerosis. The investigators will identify Treg molecular markers and changes in function in patients with relapse remitting multiple sclerosis (RRMS). The investigators plan to study T regulatory immune cells in the blood of RRMS patients and control subjects to examine how Treg immune cells' deficient function may be involved in the development of mulitple sclerosis.

DETAILED DESCRIPTION:
The study will enroll 40 RRMS patients (age 18-55, expanded disability status scale (EDSS) 0-6), and 40 age-, sex- and race-matched Healthy Controls (HCs). The study subjects will be enrolled at the Thomas Jefferson University MS clinic, which serves as a tertiary referral center.

The inclusion criteria are confirmed diagnosis of RRMS according to McDonald's diagnostic criteria12, age 18-55 inclusive, extended disability status score (EDSS) 1.5-5.5, and no immunomodulatory therapy at the time of the study. Treatment-free period will be at least 4 weeks for IV Methylprednisolone, Interferon-beta, Glatiramer acetate, Fingolimod, Tecfidera and Natalizumab. Patients previously treated with immunosuppressive therapies, including Azathioprine, Methotrexate, Mitoxantrone and Cyclophosphamide will not be enrolled in the study. Exclusion criteria will include concomitant infection, significant medical and psychiatric condition at the discretion of principal investigator. Pregnant women, and patients participating in other research trials will not be enrolled in this study. 40 healthy controls matched for age, sex and race with the group of RR MS patients will be enrolled in the study as a control group.

Aim 1. A. Identify the phenotype changes in CD4+CD25+CD127- nTregs in RRMS patients.

Transcriptional profiling of sorted CD4+CD25+CD127- Tregs will be performed using RNAseq in the first cohort of 10 HCs and 10 RRMS patients. CD4+CD25+CD127- Treg cells will be sorted from magnetic beads separated CD4+ cells. cDNA will be generated using the SMART-Seq v4 Ultra Low Input RNA Kit for Sequencing. The detection of differentially expressed genes between RRMS patients and HC-derived Treg cells will permit the functional characterization of Treg cells in RRMS. The RNA seq experiments and data analysis will be performed by Dr. Paolo Fortina and Dr. Adam Ertel at TJU Sidney Kimmel Cancer Center. The differential gene expression in RRMS Tregs identified by RNAseq will be confirmed via RT-PCR and western blotting.

Flow cytometry studies using the peripheral blood mononuclear cell (PBMC) samples from the second cohort of HCs and RRMS patients (10 donors in each group) will be used to determine changes in the expression of the Treg protein markers in RRMS patients. Individual Treg markers confer specific mechanisms of suppression. For the comprehensive Treg phenotypic profiling, the investigatorswill determine the percentage of CTLA-4, CD39, GZB, perforin, GITR, OX40, HLADR, TNFR2, Tim-3, programmed death receptor (PD-1), and LAG3-positive cells within the CD4+CD25+CD127--gated Tregs. FOXP3, GZB and perforin expression will be determined using intracellular staining, as well as Tregs' TGF-B, IL-10 and IL-35 cytokine secretion, which may contribute to their suppressive function (2x106 PBMCs per 14 color staining).

Aim 1.B. Characterize the functional deficit of nTregs in RRMS. Functional suppression assays will compare Treg suppressive function in a third cohort of 10 HC and 10 RRMS patients.

The hypothesis is that Treg co-cultures with Teff cells from HCs will increase the concentration of TGF-B, IL-10 and IL-35 and decrease the concentrations of IFN-y and IL-17A in culture supernatants (SNs) in comparison to the suppression assays using Treg and Teff cells from RRMS patients. In order to examine the susceptibility of Teff cells in RRMS patients in comparison to HCs, the suppression assays will be performed in a cross-over design experiments:

1. RMS Tregs+RRMS Teff cells
2. HC Tregs+HC Teff cells
3. RRMS Tregs+HC Teff cells
4. HC Tregs+RRMS Teff cells

Sorted 2x104 CD4+CD25+CD127- Tregs per condition will be co-cultured with autologous Teff CFSE-stained CD4+CD25-CD127+ cells in the presence of aCD3 (0.5 ug/ml) and aCD28 (1 ug/ml) mAb and 105 irradiated antigen presenting cells (PBMCs - CD4+ cells) at 1:1 and 1:10 ratios. The investigators will measure proliferation via CFSE dilution in the Teff cells and cytokine secretion in the SNs of cell cultures to determine to what extent Treg cells from RRMS patients exhibit decreased suppression in comparison to HCs. The IFN-y, IL-17A, IL-17F, IL-21, IL-10, TGF-B and IL-4 cytokine measurements will be performed using ELISA.

Aim 1.C. Determine the effects of IL-7 on the nTregs' suppressive function in RRMS.

Since our preliminary data have identified IL-7-induced STAT5 phosphorylation and FOXP3 expression, as well as IL-7 in-vitro induced Treg proliferation, the investigators will correlate the serum IL-7 levels with the Treg numbers (% of CD4+ cells x total number of cells) and their suppressive function, and examine the effect of pre-incubation of Tregs with this cytokine to their suppressive function.

Aim 2.A. Determine the phenotype of iTreg cells in RRMS patients. Flow cytometry studies of the IL-10+CD4+ and TGF-B+CD4+ cells derived from RRMS patients and HCs will identify disease-specific phenotype of iTregs, which may reflect functional changes of iTregs in RRMS. Investigators will examine the same samples from cohort of RRMS patients and HCs enrolled in Specific Aim 1.A. Flow cytometry studies of the gated CD4+IL-10+ and CD4+TGF-B+ cells will be performed using surface marker staining for CD39, CTLA-4, PD-1, ICOS, CD46, CD49b and LAG-3 and intracellular staining for FOXP3, IL-35, GZMB, pSTAT3, the repressor of GATA-3 (ROG), the aryl hydrocarbon receptor (AhR) and c-Maf transcription factors.

Aim 2.B. Identify the mechanisms of deficient nTreg induction of iTregs in RRMS.

Suppressive assay's will be performed as described in Aim 1.B using CD4+CD25+CD127-Treg and CD4+CD25-CD127+ Teff cells derived from the fourth cohort of 10 HCs and 10 RRMS patients. After 4 days of co-culture, CD25+ Treg cells will be removed using magnetic beads, and the remaining CD4+CD25- cells will be irradiated and replated at a 1:10 ratio with autologous CD4+CD25- T cells, and stimulated by plate-immobilized aCD3 and aCD28 mAb for an additional 5 days in order to demonstrate the suppressive effect of iTregs. Cell proliferation (measured by 3[H] incorporation) and TGF-β and IL-10 secretion in the SNs will be measured to determine the iTreg suppressive function induced by CD4+CD25+CD127- Tregs in the effector CD4+ cells. In the second co-culture, the investigators will also examine to what extent the iTreg induction is mediated via cell-to-cell contact (blocked by a permeable membrane) or by soluble cytokines (blocked by aIL-10, aTGF-B or aIL-4 mAb).

Aim 2.C. Characterize the effect of the iTreg-produced immunoregulatory cytokines on the reconstitution of immune tolerance.

Investigators will measure the IFN-y, IL-17A, IL-17F, IL-21, IL-22, IL-9, and IL-10, TGF-B and IL-35 levels in the SNs of the above co-cultures of iTregs and CD4+ cell derived from RRMS patients and HCs at 48 h. The investigators will measure the expression of the MHC class I and II, CD80, CD86, CD40 and CD58 in the remaining PBMC samples obtained in Specific Aim 2B in 10 HCs and 10 RRMS patients in CD19+-gated B cells, CD14+-gated monocytes, and CD1c-gated DCs using flow cytometry, as reported in our previous study 43. The investigators will examine to what extent iTreg numbers and iTregs' IL-10 and TGF-B production, as well as IL-10 and TGF-B serum levels correlate with the inhibition of MHC and costimulatory molecules' expression in B cells, monocytes and DCs in HCs and RRMS patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of RRMS according to McDonald's diagnostic criteria
* Age 18-55
* Extended disability status score (EDSS) 1.5-5.5
* No immunomodulatory therapy at the time of the study. (Treatment-free period will be at least 4 weeks for IV Methylprednisolone, Interferon-beta, Glatiramer acetate, Fingolimod, Tecfidera and Natalizumab. Patients previously treated with immunosuppressive therapies, including Azathioprine, Methotrexate, Mitoxantrone and Cyclophosphamide will not be enrolled in the study.)

Exclusion Criteria:

* Concomitant infection
* Significant medical and psychiatric condition at the discretion of principal investigator
* Pregnant women
* Patients participating in other research trials

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 Patients with relapse remitting multiple sclerosis (RRMS), 40 Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Characterize natural (n) Tregs' functional deficit in RRMS | Baseline
  Functional suppression assays will compare Treg suppressive function in a third cohort of 10 HC and 10 RRMS patients.
Identify the role of inducible (i) Treg cells in maintaining the immunological tolerance in RRMS | Baseline

SECONDARY OUTCOMES:
Identify the phenotype changes in CD4+CD25+CD127 nTregs in RRMS patients | Baseline
  Transcriptional profiling of sorted CD4+CD25+CD127- Tregs will be performed using RNAseq in the first cohort of 10 HCs and 10 RRMS patients.
Characterize functional deficits of nTregs in RRMS | Baseline
  Functional suppression assays will compare Treg suppressive function in a third cohort of 10 HC and 10 RRMS patients.
Determine the effects of hemostatic cytokines on the nTregs' suppressive function in RRMS | Baseline
Determine the phenotype of iTreg cells in RRMS | Baseline
  Flow cytometry studies of the IL-10+CD4+ and TGF-B+CD4+ cells derived from RRMS patients and HCs will identify disease-specific phenotype of iTregs, which may reflect functional changes of iTregs in RRMS.
Identify the mechanisms of deficient nTreg induction of iTregs in RRMS | Baseline
  We will perform the suppressive assay using CD4+CD25+CD127-Treg and CD4+CD25-CD127+ Teff cells derived from the fourth cohort of 10 HCs and 10 RRMS patients.
Characterize the effect of the iTreg-produced immunoregulatory cytokines on the reconstitution of immune tolerance | Baseline
  We will measure the IFN-y, IL-17A, IL-17F, IL-21, IL-22, IL-9, and IL-10, TGF-B and IL-35 levels in the SNs of the above co-cultures of iTregs and CD4+ cell derived from RRMS patients and HCs at 48 h.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States